CLINICAL TRIAL: NCT03262493
Title: Use of Feeding Tube Attachment Device Versus Conventional Fixation and Its Impact on Accidental Exit of Enteral Feeding Tubes: Randomized Clinical Trial
Brief Title: Feeding Tube Attachment Device Versus Conventional Fixation and Its Impact on Accidental Exit of Enteral Feeding Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 170217
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2017-08

CONDITIONS: Adult; Enteral Nutrition; Tube Feeding
Keywords: intubation, gastrointestinal; nursing; clinical trial; enteral nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): It consists of the use of the feeding tube attachment device (FTAD) to fix the enteral probe.
  Interventions: Device: Interventional Group
- Conventional Group (No Intervention): It consists of the fixation of the enteral probe with adhesive tape of the micropore type and plaster.

INTERVENTIONS:
Device: Interventional Group — Use of the feeding tube attachment device (FTAD).
  Arms: Interventional Group

SUMMARY:
Enteral nutritional therapy, fed through the gastrointestinal tract via a catheter, tube, catheter, or stoma, delivers the nutrients distally to the oral cavity and may reduce intrahospital malnutrition. Enteral probes are inserted, at the bedside, through the nose or mouth into the stomach or duodenum. Among the main complications of the use enteral probes, we can mention: displacement of the probe and administration of diet in the respiratory tract or microaspirations. To prevent displacement, enteral probes are attached to the skin on the nose or forehead by the use of micropore-type adhesive. In the probe the adhesive tape is put in the form of "tie" and again fixed to the nose of the patient. The enteral probes displacement rates with this technique are around 62%; in addition, the adhesive tape can cause discomfort, nasal necrosis, skin lesions and skin sensitivity reactions to the patient. More recently the nasal bridle, an anchor of the enteral feeding tube located around the nasal septum or nasal septum, has been described as more effective in securing enteral probes position over traditional tape attachment, but is not available in our environment. In Brazil, the feeding tube attachment device (FTAD) is available. Until now, the performance of FTAD in relation to enteral probe safety and accidental exit rates has not been described in the literature. Material's FTAD is composed of a layer of hydrocolloid that is adhered to the skin on the back of the nose and a polyurethane clamp that secures the enteral probe. Thus, there was a need to evaluate the actual success in using the traditional mode of probe attachment. It should be noted that very little scientific evidence is available in the literature on such care, and this is due to the lack of well-designed studies on the subject.

DETAILED DESCRIPTION:
Patients will be randomly assigned to the intervention group consisting of the use of the feeding tube attachment device (FTAD) or the control group that will use the conventional method of attachment with micropore adhesive tape and tape . The data will be compared by Student's t test or Mann-Whitney and Pearson's chi-square, according to their distribution. The project was approved by the Ethics and Research Committee of the Hospital de Clínicas de Porto Alegre. Daily will be accessed through the diet map, available in the hospital application, patients who are in use enteral nutrition. These data will be tabulated in the screening worksheet, those who meet the eligibility criteria will be invited to participate in the study and requested the reading and signing of the informed consent by the patient or guardian. The study investigator will inform the allocation group to the guest patient.By means of a structured questionnaire, socio demographic and clinical information will be collected: age, gender, reason for current hospitalization, comorbidities and information related to enteral probe (type of probe, place and date of insertion, number of medications in use via enteral probe, type and the date of the last fixation change).

Traditional fixation with micropore and plaster is routinely performed by the nursing staff every 24 hours or whenever necessary. The procedure will be performed as described in the study protocol (item 1.1).

The feeding tube attachment device (FTAD) contains a layer of hydrocolloid that will attach to the skin and a clamping clamp around the probe. The placement of the catheter fixation device will be performed by the research nurses, these will be previously trained by the manufacturer of the material. The fixing procedure is described in item 1.2.

Patients included will be evaluated daily for study outcomes up to the suspension of enteral nutrition prescription, hospital discharge, death or up to 35 days of follow-up. Patients starting enteral probe use on Saturday and Sunday can be up to 48 hours with the traditional method of fixation and later will be randomized to the intervention or control group.

1.1 Control Group After inclusion in the study, initial evaluation and information to the patient, the attending nurse will follow up on the exchange of the traditional enteral probe fixation device that occurs according to the standard operating protocol in the institution that recommends micropore fixation according to the "tie" technique and exchange Every 24 hours and whenever it is loose or with presence of dirt.

1.2 Intervention Group

After inclusion in the study and the initial evaluation, the patient will be informed of the intervention to be submitted. The care nurse will place the catheter fixation device, which according to the manufacturer, should follow the following instructions:

* Wash the patient's nose with soap and water that does not release residue;
* Rinse vigorously and dry thoroughly.
* Remove the paper that isolates the adhesive barrier (step 1);
* Position the device so that the fastener is approximately 1 cm below the tip of the nose. Apply the barrier to the patient's nose, pressing the barrier surface gently against the skin for 60 seconds (step 2);
* Fasten the feeding probe, closing the clamp around it, and firmly tighten the arms to fully engage the serrated teeth (step 3);
* To remove, raise clamp. Place the tip of one finger over the ledge on the opposite arm and turn the arm to open (step 4).

The exchange of the device should be every 7 days, in the presence of dirt or if material deterioration occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized in the clinic unit care: 6 sul e 7 norte
* Use of enteral nutrition in open system

Exclusion Criteria:

* Use of enteral nutrition by gastrostomy or jejunostomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of accidental enteral probes exit per patient | Thirty fifth day
  Will be accessed by the patient's chart

SECONDARY OUTCOMES:
Reasons for the accidental enteral probes exit per patient and / or reintegration of enteral probes between the groups | Thirty fifth day
  Will be accessed by the patient's chart
Administrated enteral nutrition volume per patient | Thirty fifth day
  The volume of enteral nutrition received will be accessed by the patient's chart
Time of fasting or delay in the use of enteral probes between groups | Thirty fifth day
  Time of fasting will be accessed by the patient's chart

CONTACTS AND LOCATIONS:
Overall Officials: Michelli S de Assis, Doctorate, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Michelli Cristina Silva de Assis, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided